CLINICAL TRIAL: NCT02118493
Title: Endo-biliary Laser Excision of Biliary Stenoses: Initial Experience and Feasibility
Brief Title: Endo-biliary Laser Excision of Biliary Stenoses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol has been withdrawn for re-evaluation.
Sponsor: University of Florida (Other)
Collaborators: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400129
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Biliary Tract Disease; Bile Duct Obstruction
Keywords: Benign Biliary Stenosis; Laser Excision
MeSH Terms: conditions — Biliary Tract Diseases; Cholestasis | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benign Biliary Stenosis, Laser (Experimental): Subjects that undergo the experimental intervention, that being single use of a laser excision catheter.
  Interventions: Device: Benign Biliary Stenosis, Laser

INTERVENTIONS:
Device: Benign Biliary Stenosis, Laser — Single use of laser to attempt excision of biliary ductal tissue causing stenosis.
  Other Names: Spectranetics Turbo-Tandem Laser Guide Catheter with Laser Atherectomy Catheter; Spectranetics CVX-300 Excimer Laser System

SUMMARY:
The biliary system normally empties into the intestines, however, some patients have biliary system narrow areas ("stenosis") that prevent the bile to drain normally. These may be related to an underlying disease or previous surgery. Patients with this problem usually require tubes to be inserted into the biliary system to drain bile into a bag outside of their body, impacting their quality of life.

The purpose of this research study is to use a laser device to try to re-open the biliary drainage system.

DETAILED DESCRIPTION:
The current preferred minimally invasive treatment for surgically related or in-situ benign biliary stenosis (BBS) involves open surgical revision, endoscopic retrograde cholangiographic (ERCP) or percutaneous transhepatic cholangiographic (PTC) balloon angioplasty and/or stent/biliary catheter placement. Unfortunately, most patients are poor open surgical operative candidates. Although ERCP is the preferred secondary approach, anatomical restrictions often require PTC. Additionally, previously placed biliary stents/catheters have poor long term patency and require routine exchange every 3-6 months. The vast majority of surgically related BBS patients are non-operative candidates for surgical revision of their BBS, and do not have favorable anatomy for ERCP access. For patients who have failed aggressive PTC balloon angioplasty of their stenoses, treatment consists of indefinite biliary catheter exchanges every 3 months. Lifelong biliary catheter dependence severely impacts the quality of life in an otherwise healthy patient with no additional evidence of their initial disease process.

A potential long-term therapy to alleviate BBS that has not been explored is the use of laser excision of the fibrotic tissue responsible for these stenoses. Therapeutic applications of lasers in medicine is not a novel concept. Its use has been well documented in the urologic tract to ablate tissue (benign prostatic hypertrophy) and renal stones. Recent laser therapeutic use in the biliary tract to dissolve gallstones has been described. The laser excision of BBS has potential to provide long term alleviation of BBS. The primary endpoint of this feasibility study is to assess the safety and initial efficacy of BBS laser excision.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed benign biliary stenosis
* Initial total serum bilirubin > 1.9 mg/dL
* Subjects currently having an internal/external percutaneous biliary drain
* Subjects that have failed at least 3 separate biliary stenosis balloon angioplasties and are deemed non-surgical candidates by the transplant and/or pancreaticobiliary surgical services at the University of Florida

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients free of post-interventional complications after use of the endo-biliary laser. | up to 100 weeks
  Patients will be assessed for safety after the endo-biliary laser use. Specifically, intraprocedural, immediate post-procedural (up to 4 hours), phone conversation 1 week post-procedure, and regularly scheduled 4 week post-procedure follow-up appointments will document the patient's tolerance of the procedure and any deviations from patients receiving biliary tube exchanges. Particular attention will be placed on regularly monitored signs/symptoms, such as cholangiographic appearance, total bilirubin, jaundice/fever/abdominal pain, etc. As each patient follows up on an ~4 week basis, any potential post-intervention complication will be documented.

SECONDARY OUTCOMES:
Technical success of endo-biliary laser excision via cholangiographic imaging. | up to 100 weeks
  Intraprocedural ability to excise fibrotic biliary tissue with the laser will be assessed by comparing pre- and immediately post-cholangiographic imaging.
Number of patients able to have internal-external biliary drainage catheters removed after endo-biliary laser excision. | up to 100 weeks
  Although this study is not powered to truly measure efficacy of this intervention, the investigators will monitor patient's for possible removal of required internal-external biliary drainage after the laser intervention. This will be monitored by 1) post-intervention follow-up cholangiograms 2) capping of the internal-external biliary drainage tube while monitoring patient symptoms and total bilirubin level and 3) possible removal of internal-external biliary tube post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Beau Toskich, MD, Principal Investigator — University of Florida Dept of Interventional Radiology

REFERENCES:
- [Background] Laasch HU, Martin DF. Management of benign biliary strictures. Cardiovasc Intervent Radiol. 2002 Nov-Dec;25(6):457-66. doi: 10.1007/s00270-002-1888-y. Epub 2002 Oct 24. PMID 12391514
- [Background] Shimada H, Endo I, Shimada K, Matsuyama R, Kobayashi N, Kubota K. The current diagnosis and treatment of benign biliary stricture. Surg Today. 2012 Dec;42(12):1143-53. doi: 10.1007/s00595-012-0333-3. Epub 2012 Sep 22. PMID 23001533
- [Background] Garcia-Cano J. Endoscopic management of benign biliary strictures. Curr Gastroenterol Rep. 2013 Aug;15(8):336. doi: 10.1007/s11894-013-0336-2. PMID 23857116
- [Background] Zarrabi A, Gross AJ. The evolution of lasers in urology. Ther Adv Urol. 2011 Apr;3(2):81-9. doi: 10.1177/1756287211400494. PMID 21869908
- [Background] Peng Q, Juzeniene A, Chen J, et al. Lasers in medicine. Reports Prog Phys. 2008;71(5):056701. doi:10.1088/0034-4885/71/5/056701.
- [Background] Kow AW, Wang B, Wong D, Sundeep PJ, Chan CY, Ho CK, Liau KH. Using percutaneous transhepatic cholangioscopic lithotripsy for intrahepatic calculus in hostile abdomen. Surgeon. 2011 Apr;9(2):88-94. doi: 10.1016/j.surge.2010.08.002. PMID 21342673
- [Background] Rimon U, Kleinmann N, Bensaid P, Golan G, Garniek A, Khaitovich B, Winkler H. Percutaneous transhepatic endoscopic holmium laser lithotripsy for intrahepatic and choledochal biliary stones. Cardiovasc Intervent Radiol. 2011 Dec;34(6):1262-6. doi: 10.1007/s00270-010-0058-x. Epub 2010 Dec 16. PMID 21161660
- [Background] Shammas NW, Shammas GA, Hafez A, Kelly R, Reynolds E, Shammas AN. Safety and One-Year revascularization outcome of excimer laser ablation therapy in treating in-stent restenosis of femoropopliteal arteries: A retrospective review from a single center. Cardiovasc Revasc Med. 2012 Nov-Dec;13(6):341-4. doi: 10.1016/j.carrev.2012.08.012. Epub 2012 Oct 6. PMID 23043953
- [Background] Steinkamp HJ, Wissgott C, Rademaker J, Scheinert D, Werk M, Settmacher U, Felix R. Short (1-10 cm) superficial femoral artery occlusions: results of treatment with excimer laser angioplasty. Cardiovasc Intervent Radiol. 2002 Sep-Oct;25(5):388-96. doi: 10.1007/s00270-002-1864-6. Epub 2002 Jun 4. PMID 12042997
- [Background] Karaca I, Ilkay E, Akbulut M, Yavuzkir M. Treatment of in-stent restenosis with excimer laser coronary angioplasty. Jpn Heart J. 2003 Mar;44(2):179-86. doi: 10.1536/jhj.44.179. PMID 12718480
- [Background] Kuo WT, Cupp JS. The excimer laser sheath technique for embedded inferior vena cava filter removal. J Vasc Interv Radiol. 2010 Dec;21(12):1896-9. doi: 10.1016/j.jvir.2010.08.013. Epub 2010 Nov 3. PMID 21050774
- [Background] Dave RM, Patlola R, Kollmeyer K, Bunch F, Weinstock BS, Dippel E, Jaff MR, Popma J, Weissman N; CELLO Investigators. Excimer laser recanalization of femoropopliteal lesions and 1-year patency: results of the CELLO registry. J Endovasc Ther. 2009 Dec;16(6):665-75. doi: 10.1583/09-2781.1. PMID 19995111
- [Background] Dachman AH, McGehee JA, Beam TE, Venbrux AC, Hoyt RF, Burris JA. Animal model for fluoroscopically guided laser application in the biliary tree. Radiology. 1990 Mar;174(3 Pt 2):1021-5. doi: 10.1148/radiology.174.3.174-3-1021. PMID 2305083